CLINICAL TRIAL: NCT03358134
Title: Mechanism of Action Study of Anti-IL17 Treatment in Spondyloarthritis: Impact on Cellular and Molecular Pathways of Synovial Inflammation and Tissue Remodeling
Brief Title: Mechanism of Action of Anti-IL17 Therapy in Peripheral Spondyloarthritis
Acronym: MoA aIL-17
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, D.L.P. Baeten, Professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AMC__45246_MoA_aIL17; 2013-002709-79 (EudraCT Number)
Record Dates: First submitted 2014-02-12; First posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Spondylarthropathies
Keywords: Peripheral Spondylarthropathies; Psoriatic arthritis; Reactive arthritis
MeSH Terms: conditions — Spondylarthropathies; Arthritis, Psoriatic; Arthritis, Reactive | interventions — secukinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Secukinumab (Experimental): All patients will be treated with active treatment. (anti-IL17)
  Interventions: Drug: Secukinumab

INTERVENTIONS:
Drug: Secukinumab — anti IL17 therapy (subcutaneous)
  Other Names: AIN457

SUMMARY:
The purpose of this study is to determine the mechanism of action on target tissue level of anti Interleukine-17 (anti-IL-17) an therapy in peripheral spondyloarthritis.

Patients will be treated with anti-IL-17 therapy (secukinumab) for 12 weeks and with a 2 year extension period thereafter.

At week 0 and 12 peripheral blood, synovial tissue and skin will be analysed with different techniques, including immunohistochemistry, RNA analysis and tissue culture to assess the effect of the therapy on inflammatory pathways.

DETAILED DESCRIPTION:
Background of the study:

Spondyloarthritis is the second most frequent form of chronic inflammatory arthritis with a prevalence of 0.5%. It effects mainly young adults and leads to major functional handicap due to inflammation of axial and peripheral joints as well as progressive ankylosis and structural damage.

In the late nineties Tumor Necrosis Factor (TNF) blockade was introduced as a successful treatment, but: only 50% responds well and tolerates, a-TNF does not halt the structural damage and TNF blockade does not induce long lasting remission as almost all patients relapse within a few weeks after interruption of the treatment. There is thus a high unmet need for alternatives.

The rationale for anti-IL17 therapy is based on various auto-inflammatory and auto immune models, preliminary efficacy data in psoriasis and Rheumatoid arthritis (RA) and an association of SpA with Interleukin 23 Receptor (IL23R) single nucleotide polymorphism (SNP).

Efficacy data on anti-IL17 shows that it is a highly effective treatment for signs and symptoms in SpA, moreover sub-analysis of the anti-TNF naïve patients shows the same trend.

Objective of the study:

To assess molecular and cellular effects of the treatment on the synovium.

Secondary:

To compare which molecular and cellular disease pathways are affected by IL-17 blockade and not by TNF blockade and thereby identify molecular biomarkers which may help to determine which patients may benefit form this treatment in comparison with anti-TNF treatment.

To assess wether AIN457 silences vessel wall inflammation (by means of 18F-FDG PET(positron emission tomography)/CT of the carotic arteries and aorta.

Study design:

Single centre, 12-week open label study in subjects with clinically active peripheral spondylarthritis, with open label extension up to 2 years. Synovial biopsies and 18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose (18F FDG) PET/CT of the aorta and carotid arteries will be obtained from patients before and after 12 weeks of treatment with secukinumab.

Study population:

Patients with a diagnosis of spondyloarthritis according to the European Spondyloarthropathy Study Group (ESSG) or Assess Spondyloarthritis to international Society (ASAS) criteria with at least one swollen knee or ankle joint.

Intervention :

Secukinumab (AIN457) by subcutaneous injections (weekly for the first 4 weeks and every 4 weeks thereafter).

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant/non-lactating females age 18-70
* Diagnosis of SpA according to ESSG criteria and/or ASAS criteria
* Active disease defined by ≥1 swollen and ≥ 1 tender joint, and at least 1 swollen knee or ankle joint at baseline

Exclusion Criteria:

* Evidence for infectious or malignant process (on chest X ray/MRI etc)
* Patients taking opioid analgetics
* Previous IL-17 therapy exposure
* Previous use of cell-depleting therapies, biological immunomodulators (except for TNF blockade , as 25% may have been previously treated with 1 TNF blocking agent)
* Significant medical problems or diseases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-03; Primary Completion 2017-07 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Biological changes induced by therapy on target tissue (synovium) | week 0 and week 12
  Molecular changes of the synovium as measured by expression of several cytokines/chemokines by quantitative polymerase chain reaction (qPCR) as measured by a change in cytokine expression between baseline and week 12.
Changes of cellular infiltrate in the target tissue (synovium) | week 0 and week 12
  Changes in cell count measured by immunohistochemistry (on a 0-4 semi-quantitative analysis scale)

SECONDARY OUTCOMES:
Adverse events | between day0 and 2 yrs of treatment
  Number of patients with adverse events as a measure of safety and tolerability
Vessel wall inflammation | week 0 and week 12
  Changes in Fludeoxyglucose (FDG18) PET/CT uptake in the vessel walls of the carotic arteries and aorta as measured by CT values

CONTACTS AND LOCATIONS:
Overall Officials: dominique LP Baeten, MD PhD prof., Principal Investigator — AIDS Malignancy Consortium
Locations (1):
- Academic Medical Center Amsterdam, Amsterdam, North Holland, Netherlands